CLINICAL TRIAL: NCT03670849
Title: Ultrasound Augmentation of Stereoscopic and Conventional Video for Laparoscopic Surgeries
Brief Title: Image Fusion in the OR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raj Shekhar (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); IGI Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Raj Shekhar, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00003344; 2R42CA192504 (NIH)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Laparoscopic Cholecystectomy; Liver Ablation
Keywords: Laparoscopic Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients using LapAR system (Experimental)
  Interventions: Device: LapAR

INTERVENTIONS:
Device: LapAR — LapAR system will map (transform) the live LUS image in the reference frame of the laparoscopic camera, and fuse it with the live laparoscopic video in real time. For thermal ablations that involve a needle, we also track the needle and overlay its path on the AR view.

SUMMARY:
The objective of this study is to test the technical feasibility of LapAR visualization system for guiding laparoscopic surgeries and to gather clinical feedback on the use of this tool.

DETAILED DESCRIPTION:
Surgeons use real-time video generated by a laparoscope to visualize the operative field when performing laparoscopic procedures. An inability to see beneath organ surfaces is a limitation of the current visualization technology. Surgeons additionally use laparoscopic ultrasound to see beneath organ surfaces, but also need to mentally correlate the ultrasound image with the video of the operative field. This process is difficult, subjective, and variable with expertise, and discourages the use of ultrasound.

We have developed a method to combine live laparoscopic video and laparoscopic ultrasound images to present fused multimodality images on a single display, eliminating the need for mental image correlation. Specifically, the image fusion method, called laparoscopic augmented reality (LapAR), augments the laparoscopic video with ultrasound data when required by surgeons. For ablations, we further track the needle and overlay its path on the AR view for precise needle placement. This study is designed to test this minimal-risk capability in patients referred for relevant laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Referred for laparoscopic cholecystectomy or liver ablation
2. Clinical indication for the use of laparoscopic ultrasound
3. Patient or an authorized guardian provides written consent

Exclusion Criteria:

Patients with pacemaker or any other ICD (intra-cardiac device) which may interfere with electromagnetic tracking

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Usability | post surgery, an expected average of 5 minutes
  The ease of use of the LapAR system will be evaluated by the surgeon
System set-up time | before surgery, an expected average of 15 min

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States